CLINICAL TRIAL: NCT00120523
Title: Five-Year Safety Study of Pimecrolimus Cream 1% in Infants 3 to Less Than 12 Months of Age With Mild to Moderate Atopic Dermatitis
Brief Title: 5-Year Safety Study of Pimecrolimus Cream 1% in Infants 3 - 12 Months of Age With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASM981C2306
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2016-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, children, infants, pimecrolimus
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Active Comparator): Topical corticosteroids
  Interventions: Drug: Topical corticosteroids

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel
  Arms: 1
Drug: Topical corticosteroids — TCS
  Arms: 2

SUMMARY:
The primary purpose of this study is to investigate the safety of pimecrolimus cream 1% in the long-term treatment (up to 5 years) of atopic dermatitis (eczema) in patients less than 12 months of age compared to topical corticosteroids (TCS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to < 12 months
* Diagnosis of AD fulfilling the diagnostic criteria of Seymour
* AD affecting at least 5% total body surface area
* Investigator's Global Assessment (IGA) score of 2 or 3, corresponding to mild-to-moderate disease at baseline
* Informed consent

Exclusion Criteria:

* Phototherapy, systemic therapy (e.g., immunosuppressants, cytostatics), systemic corticosteroids within 4 weeks
* Topical tacrolimus or pimecrolimus within 2 weeks
* Topical therapy (e.g., tar, topical corticosteroids) within 3 days
* Immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have a history of malignant disease
* Active acute viral skin infection (e.g. herpes simplex, herpes zoster, chicken pox), and/or clinically infected AD
* Failure to thrive (e.g., weight or height/length below the 5th percentile) or developmental abnormalities such as head circumference less than 5th and more than 95th percentile
* Known hypersensitivity to any ingredient of pimecrolimus cream 1% or topical corticosteroids
* Clinical conditions other than AD that according to investigator can interfere with the evaluation

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2418 (Actual)
Dates: Start 2004-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Cholla Pediatrics, Tucson, Arizona
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Little Rock Allergy & Asthma Clinic, Little Rock, Arkansas
  - 9540 Artesia Blvd., Suite #1, Bellflower, California
  - Pediatric Care Medical Group, Inc., Huntington Beach, California
  - Longmont Clinical Research, Longmont, Colorado
  - Children's Skin Center, Miami, Florida
  - Pediatric Research Center of South Florida, Palm Beach Gardens, Florida
  - AeroAllergy Research Laboratories of Savanah, Inc., Savannah, Georgia
  - The Pediatric Center, Stone Mountain, Georgia
  - Wayne State University Dermatology, Detroit, Michigan
  - Michigan State University - Kalamazoo Center for Med Studies, Kalamazoo, Michigan
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - SMDC Health System, Duluth, Minnesota
  - Dermatology Center for Children, Minneapolis, Minnesota
  - University of Minnesota - Dept. of Dermatology, Minneapolis, Minnesota
  - Radiant Research, Bridgeton, Missouri
  - Dermatology Associates of Rochester, P.C., Rochester, New York
  - Capitol Pediatrics & Adolescent Center, Raleigh, North Carolina
  - Dermatology Research Associates, Cincinnati, Ohio
  - Ohio Pediatrics, Inc., Huber Heights, Ohio
  - The Portland Clinic, Beaverton, Oregon
  - Calcagno Research and Development, Gresham, Oregon
  - Allergy & Asthma Consultants, LLP, Charleston, South Carolina
  - Allergic Disease and Asthma Center, Greenville, South Carolina
  - University of Tennessee - Dept. of Pediatrics, Memphis, Tennessee
  - Suzanne Bruce& Associates, PA, Houston, Texas
  - Grand Parkway Pediatrics, Sugar Land, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Novartis, Investigative Site, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sigurgeirsson B, Boznanski A, Todd G, Vertruyen A, Schuttelaar ML, Zhu X, Schauer U, Qaqundah P, Poulin Y, Kristjansson S, von Berg A, Nieto A, Boguniewicz M, Paller AS, Dakovic R, Ring J, Luger T. Safety and efficacy of pimecrolimus in atopic dermatitis: a 5-year randomized trial. Pediatrics. 2015 Apr;135(4):597-606. doi: 10.1542/peds.2014-1990. Epub 2015 Mar 23. PMID 25802354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled into the study on 05 Apr 2004, last patient completed on 04 Oct 2010.
Groups:
- Pimecrolimus: 1% cream was supplied in 50 g tubes by the sponsor. Elidel was to be applied as a thin layer to the affected skin b.i.d., and rubbed in gently and completely by the primary caregiver
- Topical Corticosteroids: Low or medium potency (low potency, e.g. Hydrocortisone acetate; or medium potency, e.g.
  Fluticasone propionate)TCS supplied locally were to be used according to the country's label as study medication for patients randomized to TCS group. Topical corticosteroids were to be applied as a thin layer to the affected skin only and rubbed in gently.
Period: Treatment Period
Arm/Group | Pimecrolimus | Topical Corticosteroids
Started | 1205 | 1213
Completed | 836 | 874
Not Completed | 369 | 339
Period: Follow-Up Period
Arm/Group | Pimecrolimus | Topical Corticosteroids
Started | 120 (Patients discontinued due to lost to follow-up or who withdrew consent were not part of this period.) | 70 (Patients discontinued due to lost to follow-up or who withdrew consent were not part of this period.)
Completed | 90 | 46
Not Completed | 30 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimecrolimus | Topical Corticosteroids | Total
Number analyzed (Participants) | 1205 | 1213 | 2418
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1205 | 1213 | 2418
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.1 (2.71) | 7.1 (2.66) | 7.1 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 471 | 932
  Male | 744 | 742 | 1486
Region of Enrollment [Number; unit: participants]
  United States | 106 | 110 | 216
  Germany | 130 | 131 | 261
  Argentina | 40 | 40 | 80
  Belgium | 20 | 16 | 36
  Canada | 52 | 64 | 116
  Chile | 25 | 22 | 47
  China | 60 | 59 | 119
  Colombia | 48 | 52 | 100
  Czech Republic | 26 | 23 | 49
  Ecuador | 15 | 13 | 28
  Spain | 51 | 48 | 99
  United Kingdom | 32 | 27 | 59
  Greece | 19 | 16 | 35
  Guatemala | 53 | 56 | 109
  Hong Kong | 5 | 4 | 9
  Hungary | 39 | 40 | 79
  Iceland | 97 | 98 | 195
  Netherlands | 51 | 55 | 106
  Peru | 55 | 51 | 106
  Poland | 37 | 36 | 73
  Portugal | 5 | 5 | 10
  Russian Federation | 54 | 53 | 107
  Singapore | 12 | 13 | 25
  Sweden | 29 | 29 | 58
  Turkey | 26 | 28 | 54
  Taiwan | 30 | 30 | 60
  Venezuela | 39 | 39 | 78
  South Africa | 49 | 55 | 104

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed by Adverse Events
Description: crude incidence of adverse events of primary interest and most frequent adverse events (greater than or equal to 5% crude incidence in either treatment group) in the treatment period
Time Frame: throughout the 5-year study
Population: complete safety/ITT population of experimental and control
Measure: Number; unit: percentage of participants
Groups:
- Pimecrolimus: Pimecrolimus 1% cream was supplied in 50 g tubes by the sponsor. Elidel was to be applied as a thin layer to the affected skin b.i.d., and rubbed in gently and completely by the primary caregiver
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1205 | 1213
percentage of participants
  Acute tonsillitis | 8.6 | 7.8
  Allergy to arthropod bite | 5.9 | 4.9
  Arthropod bite | 7.1 | 8.8
  Asthma | 15.1 | 14.6
  Bronchiolitis | 5.4 | 5.7
  Bronchitis | 36.3 | 33.8
  Bronchospasm | 5.2 | 6.7
  Conjunctivitis | 16.5 | 16.2
  Conjunctivitis allergic | 5.0 | 6.3
  Constipation | 6.9 | 6.7
  Cough | 29.9 | 30.4
  Dermatitis diaper | 12.5 | 11.3
  Diarrhoea | 31.9 | 31.4
  Eczema infected | 7.4 | 4.5
  Eye infection | 0.3 | 0.3
  Food allergy | 7.4 | 6.0
  Gastroenteritis | 28.2 | 27.1
  Gastroenteritis viral | 6.1 | 5.2
  Heat rash | 5.5 | 4.8
  Hypersensitivity | 2.0 | 1.9
  Immunisation reaction | 6.5 | 5.5
  Impetigo | 11.9 | 10.4
  Influenza | 6.9 | 5.7
  Influenza like illness | 16.7 | 16.6
  Laryngitis | 5.4 | 4.9
  Lower respiratory tract infection | 3.7 | 4.5
  Molluscum contagiosum | 9.0 | 8.2
  Nasopharyngitis | 59.0 | 58.9
  Otitis media | 34.7 | 31.7
  Otitis media acute | 12.4 | 11.6
  Pharyngitis | 17.8 | 19.0
  Pneumonia | 11.0 | 10.8
  Pyrexia | 48.9 | 49.9
  Rhinitis | 13.9 | 13.4
  Rhinitis allergic | 13.2 | 12.7
  Rhinorrhoea | 6.8 | 6.8
  Sinusitis | 7.6 | 8.1
  Teething | 14.9 | 14.9
  Tonsillitis | 16.9 | 16.5
  Upper respiratory tract infection | 32.0 | 31.2
  Urinary tract infection | 4.3 | 5.2
  Urticaria | 9.5 | 10.6
  Varicella | 25.4 | 23.4
  Viral rash | 3.0 | 4.1
  Viral upper respiratory tract infection | 10.5 | 10.4
  Vomiting | 22.5 | 21.3
  Wheezing | 5.6 | 5.3

2. Primary Outcome: Growth Velocity (Height)
Time Frame: throughout the 5-year study
Population: Safety/intent-to-treat (ITT) - all randomized patients who received at least one application of study medication.Patient who do not have a baseline value are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1204 | 1208
cm
  Baseline (n=1204, n=1208) | 68.8 (5.26) | 68.8 (5.14)
  Week 6 (n=1144, n=1141) | 71.3 (4.82) | 71.3 (4.76)
  Week 26 (n=1092, n=1114) | 77.0 (4.37) | 76.9 (4.46)
  Week 52 (n=999, n=1052) | 83.1 (4.23) | 83.1 (4.30)
  Week 104 (n=924, n=975) | 93.0 (4.31) | 92.9 (4.30)
  Week 156 (n=871, n=919) | 100.5 (4.70) | 100.6 (4.72)
  Week 208 (n=843, n=869) | 107.7 (5.46) | 107.8 (5.25)
  Week 260 (n=833, n=871) | 114.4 (5.26) | 114.5 (5.90)

3. Primary Outcome: Growth Velocity (Weight)
Time Frame: throughout the 5-year study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1203 | 1213
kg
  Baseline (n=1203, n=1213) | 8.2 (1.51) | 8.2 (1.51)
  Week 6 (n=1144, n=1144) | 8.8 (1.45) | 8.7 (1.41)
  Week 26 (n=1093, n=1114) | 10.2 (1.43) | 10.1 (1.39)
  Week 52 (n=1003, n=1054) | 11.6 (1.52) | 11.6 (1.54)
  Week 104 (n=928, n=978) | 14.1 (1.90) | 14.1 (1.83)
  Week 156 (n=873, n=924) | 16.3 (2.32) | 16.3 (2.29)
  Week 208 (n=843, n=870) | 18.6 (2.80) | 18.7 (2.88)
  Week 260 (n=833, n=871) | 21.1 (3.51) | 21.4 (3.70)

4. Secondary Outcome: Investigator's Global Assessment (to Assess Disease Severity) of the Whole Body and of the Face: Treatment Success Rate
Description: IGA = Investigator's global Assessment. CI = Confidence interval for treatment success using binomial distribution: lower CI<0 is set to 0, upper CI>100 is set to 100.
  Treatment success (n): IGA score of 0 or 1 (clear or almost clear). Outcome gives percentage of patients with treatment success.
Time Frame: throughout the 5-year study
Population: Safety/intent-to-treat (ITT) - all randomized patients who received at least one application of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1205 | 1213
percentage of participants
  Overall IGA Week 6 | 61.4 [58.5 to 64.2] | 59.6 [56.8 to 62.5]
  Overall IGA Week 26 | 66.4 [63.6 to 69.2] | 74.5 [71.9 to 77.0]
  Overall IGA Week 52 | 73.9 [71.2 to 76.6] | 79.6 [77.2 to 82.1]
  Overall IGA Week 104 | 79.9 [77.3 to 82.4] | 83.4 [81.0 to 85.7]
  Overall IGA Week 156 | 81.9 [79.3 to 84.4] | 86.1 [83.9 to 88.3]
  Overall IGA Week 208 | 86.2 [83.8 to 88.5] | 88.1 [86.0 to 90.2]
  Overall IGA Week 260 | 88.7 [86.6 to 90.9] | 92.3 [90.5 to 94.1]
  Facial IGA Week 6 | 68.9 [66.3 to 71.6] | 71.0 [68.4 to 73.6]
  Facial IGA Week 26 | 79.5 [77.1 to 81.9] | 83.8 [81.6 to 86.0]
  Facial IGA Week 52 | 85.6 [83.4 to 87.7] | 88.5 [86.6 to 90.4]
  Facial IGA Week 104 | 92.1 [90.4 to 93.9] | 94.1 [92.6 to 95.6]
  Facial IGA Week 156 | 94.2 [92.6 to 95.7] | 94.3 [92.8 to 95.8]
  Facial IGA Week 208 | 96.0 [94.7 to 97.3] | 96.2 [95.0 to 97.5]
  Facial IGA Week 260 | 96.6 [95.4 to 97.9] | 97.2 [96.2 to 98.3]

5. Secondary Outcome: Body Surface Area Involved With Atopic Dermatitis
Description: TBSA = Total body surface area; percent BSA affected = (BSA affected/TBSA) x 100.
Time Frame: throughout the 5-year study
Population: Safety/intent-to-treat (ITT) - all randomized patients who received at least one application of study medication.
Measure: Mean (Standard Deviation); unit: percentage of TBSA affected
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1205 | 1213
percentage of TBSA affected
  Baseline (n=1205, n=1213) | 21.1 (16.50) | 21.3 (17.19)
  Week 6 (n=1142, n=1138) | 5.5 (8.72) | 6.0 (9.10)
  Week 26 (n=1091, n=1113) | 4.3 (8.30) | 3.7 (8.50)
  Week 52 (n=997, n=1048) | 3.5 (7.69) | 2.7 (6.27)
  Week 104 (n=922, n=975) | 2.4 (6.53) | 1.8 (5.17)
  Week 156 (n=871, n=918) | 2.0 (5.46) | 1.4 (4.65)
  Week 208 (n=843, n=868) | 1.5 (5.16) | 1.2 (4.33)
  Week 260 (n=833, n=870) | 1.1 (3.31) | 0.9 (3.69)

6. Secondary Outcome: Parent's Index of Quality of Life - Atopic Dermatitis (PIQoL-AD)
Description: PIQoL-AD questionnaire (28 questions) was only done in countries where validated questionnaire was available: Germany, Hungary, Netherlands, Spain, UK and US.
  For the purposes of data presentation, a "Not True" response was coded a value of zero and a "True" a value of one. The total score (i.e., sum of individual questions) was calculated; lower the score, better the QoL. Minimum score = 0; maximum score = 28. If the patient has answered ≤14 questions at a time point, then the patient's total score at the time point was set to missing.
Time Frame: throughout the 5-year study
Population: Safety/intent-to-treat (ITT) - all randomized patients who received at least one application of study medication. Patients who do not have baseline value are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 406 | 405
units on a scale
  Baseline (n=406, n=405) | 8.1 (5.04) | 8.4 (5.25)
  Week 6 (n=378, n=360) | 5.8 (4.76) | 6.0 (5.09)
  Week 26 (n=368, n=363) | 4.8 (4.73) | 5.0 (4.85)
  Week 52 (n=327, n=334) | 4.2 (4.45) | 4.4 (4.94)
  Week 104 (n=302, n=296) | 3.7 (4.69) | 3.9 (5.14)
  Week 156 (n=269, n=266) | 3.2 (4.67) | 3.4 (5.02)
  Week 208 (n=254, n=256) | 2.7 (3.93) | 3.0 (4.88)
  Week 260 (n=249, 249) | 2.1 (3.22) | 2.3 (3.80)

7. Secondary Outcome: Vital Signs and Physical Examinations: Blood Pressure (BP)
Description: Significant findings are included in the relevant medical history/current medical conditions (prior to study start) or in the AE documentation (after study start.
Time Frame: throughout the 5-year study
Population: Safety/intent-to-treat (ITT) - all randomized patients who received at least one application of study medication.Patients who do not have baseline value are excluded from analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1205 | 1213
mmHg
  Systolic BP - Baseline | 94.3 (12.40) | 94.7 (12.79)
  Systolic BP- Week 6 | 96.1 (11.70) | 96.3 (11.33)
  Systolic BP- Week 26 | 98.6 (11.46) | 98.4 (11.49)
  Systolic BP- Week 52 | 99.0 (11.33) | 99.3 (11.02)
  Systolic BP- Week 104 | 98.8 (10.01) | 97.9 (9.85)
  Systolic BP- Week 156 | 99.0 (9.47) | 98.6 (9.75)
  Systolic BP- Week 208 | 99.8 (10.10) | 99.4 (9.74)
  Systolic BP- Week 260 | 100.0 (9.51) | 100.1 (9.63)
  Diastolic BP - Baseline | 59.2 (10.40) | 59.1 (10.26)
  Diastolic BP - Week 6 | 60.4 (9.47) | 61.0 (9.59)
  Diastolic BP - Week 26 | 61.7 (9.90) | 61.6 (9.78)
  Diastolic BP - Week 52 | 61.9 (9.12) | 61.9 (9.23)
  Diastolic BP - Week 104 | 61.8 (8.14) | 61.7 (7.72)
  Diastolic BP - Week 156 | 62.0 (8.11) | 62.0 (8.29)
  Diastolic BP - Week 208 | 62.4 (8.52) | 61.8 (7.77)
  Diastolic BP - Week 260 | 61.9 (7.24) | 62.2 (7.38)

8. Primary Outcome: Potential Effect on the Developing Immune System
Description: number (%) of patients with positive antibody titers to tetanus, hepatitis B, and measles vaccines at baseline, weeks 26 (6 months), 52 (1 year), 104 (2 years), 156 (3 years), 208 (4 years) and 260 (5 years) Varicella antibody titers were measured at the above time points in US patients only.
Time Frame: throughout the 5-year study
Population: Immune system function data analyses were performed on the immunology set (774 patients). Varicella titers were assessed for USA patients only (n= 104, n=108).
Measure: Number; unit: % of patients with positive ab titer
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 383 | 391
% of patients with positive ab titer
  Tetanus Baseline | 81.8 | 85.2
  Tetanus week 26 | 89.5 | 90.4
  Tetanus week 52 | 91.9 | 94.0
  Tetanus week 104 | 91.9 | 94.7
  Tetanus week 156 | 93.5 | 92.5
  Tetanus week 208 | 89.0 | 89.5
  Tetanus week 260 | 91.1 | 88.9
  Hepatitis B Baseline | 57.5 | 53.6
  Hepatitis B week 26 | 60.7 | 58.6
  Hepatitis B week 52 | 59.0 | 58.5
  Hepatitis B week 104 | 51.5 | 51.3
  Hepatitis B week 156 | 48.5 | 45.0
  Hepatitis B week 208 | 39.7 | 38.5
  Hepatitis B week 260 | 34.6 | 38.2
  Measles Baseline | 11.4 | 14.4
  Measles week 26 | 37.4 | 31.6
  Measles week 52 | 86.3 | 86.1
  Measles week 104 | 97.3 | 97.4
  Measles week 156 | 98.5 | 97.0
  Measles week 208 | 97.8 | 95.6
  Measles week 260 | 98.9 | 96.3
  Varicella Baseline | 32.1 | 17.8
  Varicella week 26 | 46.5 | 45.2
  Varicella week 52 | 72.2 | 74.2
  Varicella week 104 | 78.4 | 88.7
  Varicella week 156 | 68.4 | 81.8
  Varicella week 208 | 86.1 | 89.4
  Varicella week 260 | 87.1 | 84.1

9. Secondary Outcome: Vital Signs and Physical Examinations: Pulse
Description: as for outcome 7
Time Frame: throughout the 5-year study
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pimecrolimus | Topical Corticosteroids
Number analyzed (Participants) | 1205 | 1213
bpm
  Baseline | 116.7 (19.43) | 116.0 (19.69)
  Week 6 | 114.2 (18.19) | 114.5 (19.45)
  Week 26 | 111.4 (18.09) | 111.7 (18.44)
  Week 52 | 107.7 (18.63) | 107.0 (17.92)
  Week 104 | 101.7 (15.97) | 101.8 (15.91)
  Week 156 | 97.4 (13.45) | 97.0 (13.72)
  Week 208 | 93.4 (12.78) | 93.4 (12.56)
  Week 260 | 90.2 (12.82) | 90.4 (12.25)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period of 5 years.
Arm/Group | Pimecrolimus | Topical Corticosteroids
Serious Adverse Events (participants affected / at risk) | 247/1205 | 210/1213
Other Adverse Events (participants affected / at risk) | 1162/1205 | 1160/1213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimecrolimus (N=1205) | Topical Corticosteroids (N=1213)
Lymphadenitis (Blood and lymphatic system disorders) | 6 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute chest syndrome (Blood and lymphatic system disorders) | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Arrhytmia (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 3
Cryptorchism (Congenital, familial and genetic disorders) | 3 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 | 0
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1
Hereditary fructose intolerance (Congenital, familial and genetic disorders) | 0 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Amblyopia (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 17 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Inguinal hernia (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 2 | 0
Intussusception (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Disbacteriosis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 3
Malaise (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Hyperplasia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Vaccination site hypersensitivity (General disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Food allergy (Immune system disorders) | 3 | 2
Anaphylactic reaction (Immune system disorders) | 3 | 1
Milk allergy (Immune system disorders) | 0 | 3
Anaphylactic shock (Immune system disorders) | 0 | 1
Antiphospholipid syndrome (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 28
Gastroenteritis (Infections and infestations) | 20 | 24
Bronchitis (Infections and infestations) | 23 | 16
Bronchopneumonia (Infections and infestations) | 9 | 18
Bronchiolitis (Infections and infestations) | 7 | 12
Gastroenteritis rotavirus (Infections and infestations) | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 9
Gastroenteritis viral (Infections and infestations) | 9 | 6
Lower respiratory tract infection (Infections and infestations) | 3 | 8
Otitis media (Infections and infestations) | 5 | 5
Pharyngitis (Infections and infestations) | 5 | 3
Croup infections (Infections and infestations) | 3 | 4
Tonsillitis (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 2 | 5
Cellulitis (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 4 | 2
Viral infection (Infections and infestations) | 4 | 2
Lobar pneumonia (Infections and infestations) | 2 | 3
Acute tonsillitis (Infections and infestations) | 4 | 0
Laryngitis (Infections and infestations) | 3 | 1
Otitis media acute (Infections and infestations) | 2 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 3
Abscess limb (Infections and infestations) | 2 | 1
Eczema infected (Infections and infestations) | 3 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 1
Gastroenteritis salmonella (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 0 | 3
Pneumonia mycoplasmal (Infections and infestations) | 0 | 3
Respiratory tract infection (Infections and infestations) | 2 | 1
Viral diarrhoea (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 1
Exanthema subitum (Infections and infestations) | 0 | 2
Gastroenteritis bacterial (Infections and infestations) | 1 | 1
Herpangina (Infections and infestations) | 0 | 2
Impetigo (Infections and infestations) | 2 | 0
Infected bites (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 1 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2
Pneumonia viral (Infections and infestations) | 1 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 0
Rotavirus infection (Infections and infestations) | 1 | 1
Subcutaneous abcess (Infections and infestations) | 2 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 2
Varicella (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Adenoiditis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Application site infection (Infections and infestations) | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bacterial rhinitis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Dysentery (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1
Gastroenteritis astroviral (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis infectious (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Kaposi's varicelliform eruption (Infections and infestations) | 1 | 0
Laryngotracheitis obstructive (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 1 | 0
Meningococcal bacteraemia (Infections and infestations) | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Naspoharyngitis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Viral skin infection (Infections and infestations) | 0 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0
Viral tracheitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 4 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Accidential drug intake by child (Injury, poisoning and procedural complications) | 0 | 1
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Rotavirus test positive (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 18 | 9
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 3
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Febrile convulsion (Nervous system disorders) | 6 | 3
Autism (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyperkinesia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 1
Tongue biting (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Autism spectrum disorder (Psychiatric disorders) | 0 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Penile adhesion (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 25 | 19
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sleep apnoe syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchial obstuction (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mouth breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Kawasaki's disease (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pimecrolimus (N=1205) | Topical Corticosteroids (N=1213)
Nasopharyngitis (Infections and infestations) | 711 | 715
Pyrexia (General disorders) | 589 | 605
Bronchitis (Infections and infestations) | 438 | 410
Otitis media (Infections and infestations) | 418 | 385
Diarrhoea (Gastrointestinal disorders) | 384 | 381
Upper respiratory tract infection (Infections and infestations) | 386 | 378
Cough (Respiratory, thoracic and mediastinal disorders) | 360 | 369
Gastroenteritis (Infections and infestations) | 340 | 329
Varicella (Infections and infestations) | 306 | 284
Vomiting (Gastrointestinal disorders) | 271 | 258
Pharyngitis (Infections and infestations) | 215 | 231
Tonsillitis (Infections and infestations) | 204 | 200
Influenza like illness (General disorders) | 201 | 201
Conjunctivitis (Eye disorders) | 199 | 197
Teething (Gastrointestinal disorders) | 179 | 181
Asthma (Respiratory, thoracic and mediastinal disorders) | 182 | 177
Rhinitis (Infections and infestations) | 168 | 163
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 159 | 154
Otitis media acute (Infections and infestations) | 150 | 141
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 151 | 137
Impetigo (Infections and infestations) | 143 | 126
Pneumonia (Infections and infestations) | 133 | 131
Viral upper respiratory tract infection (Infections and infestations) | 126 | 126
Urticaria (Skin and subcutaneous tissue disorders) | 114 | 129
Molluscum contagiosum (Infections and infestations) | 109 | 99
Acute tonsillitis (Infections and infestations) | 104 | 95
Arthropode bite (Injury, poisoning and procedural complications) | 86 | 107
Sinusitis (Infections and infestations) | 91 | 98
Constipation (Gastrointestinal disorders) | 83 | 81
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 82 | 82
Food allergy (Immune system disorders) | 89 | 73
Influenza (Infections and infestations) | 83 | 69
Immunisation reaction (Immune system disorders) | 78 | 67
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 63 | 81
Eczema infected (Infections and infestations) | 89 | 55
Conjunctivitis allergic (Eye disorders) | 60 | 76
Gastroenteritis viral (Infections and infestations) | 73 | 63
Bronchiolitis (Infections and infestations) | 65 | 69
Wheezing (Respiratory, thoracic and mediastinal disorders) | 68 | 64
Allergy to arthropod bite (Immune system disorders) | 71 | 59
Heat rash (Skin and subcutaneous tissue disorders) | 66 | 58
Laryngitis (Infections and infestations) | 65 | 59
Oral candidiasis (Infections and infestations) | 56 | 59
Urinary tract infection (Infections and infestations) | 52 | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No